CLINICAL TRIAL: NCT00266331
Title: Prospective Blinded Randomized Study; RayGel Versus Placebo-an Alternative for Skin Care During External Beam Radiation.
Brief Title: RayGel-An Alternative for Skin Care During External Beam Radiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathalie Johnson (Other)
Responsible Party: Sponsor-Investigator, Nathalie Johnson, Principal investigator, Legacy Health System
Organization: Legacy Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NW-05TJohn-01; LHS Foundation
Record Dates: First submitted 2005-12-14; First posted 2005-12-16 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Radiation skin protection
MeSH Terms: conditions — Breast Neoplasms | interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A, RayGel Topical Cream (Active Comparator): RayGel Topical Cream applied in thin layer to the area exposed to radiation 60-90 minutes prior to radiotherapy, standard skin care between treatments.
  Interventions: Drug: Reduced glutathione
- Arm B Placebo Topical Cream (Placebo Comparator): Placebo Topical Cream applied in thin layer to the area exposed to radiation 60-90 minutes prior to radiotherapy, standard skin care between treatments.

INTERVENTIONS:
Drug: Reduced glutathione
  Arms: Group A, RayGel Topical Cream

SUMMARY:
This study is for the patient with breast cancer. To take part in this study, external beam radiation therapy needs to be part of the treatment plan. Reduced glutathione, an ingredient of RayGel™, has been helpful in decreasing some radiation therapy side effects to the skin.

Reduced glutathione plays a vital role in both making DNA and cell repair. This study will measure if RayGel decreases skin reaction in breast cancer patients treated with external beam radiation therapy.

DETAILED DESCRIPTION:
RayGel versus Placebo- An Alternative for Skin Care during External Beam Radiation Therapy

RayGel is a formulation of reduced glutathione and anthocyanins extracts from various blue/purple flowering plants. Glutathione has been studied in a variety of ways in conjunction with therapies directed at cancer. It is a functional molecule, which plays a significant role in maintenance of normal cellular metabolism and regulation. Reduced glutathione plays an essential role in DNA synthesis and repair, as well as leukotriene and prostaglandin metabolism. Studies have looked at using glutathione to reduce the complication of chemotherapy such as bone pain with Taxol, and urinary effects with cyclophosphamide, and neurotoxicity with cisplatin. It has shown efficacy in these arenas.

External beam radiation is a standard part of breast conservation treatment. It reduces rates of loco regional recurrence significantly. Skin reaction of varying degrees occurs in everyone under going treatment. Occasionally, it can be so severe that the treatment schedule must be altered to allow healing. We would like to study the effect that topical RayGel may have on reducing the reaction of skin during external beam radiation therapy of the breast.

Ineligibility criteria:

1. Post mastectomy
2. Previous irradiation of the same breast
3. Pregnancy
4. Younger than 18 years of age

Contraindication:

1.Hypersensitivity

Study Design:

Prospective blinded randomized study. Enroll 150 patients.

Group A - RayGel topical cream is applied in a thin layer to the area exposed to radiation 60-90 minutes prior to radiotherapy, standard skin care between treatments.

Group B - Placebo topical cream is applied in a thin layer to the area exposed to radiation 60-90 minutes prior to radiotherapy, standard skin care between treatments.

In addition, patients with bright erythema reaction will use skin products at the discretion of the radiation oncologist.

Patients would be consented prior to start of therapy. Digital photos of the radiation area would be taken at start, ~ 5 weeks and evaluated by the radiation oncologist using the 0-6 Skin Reaction Scale. (0-no changes to 6-ulceration, hemorrhage or necrosis).

Weekly skin assessments and documentation of changes would be performed by the radiation oncology nurse and radiation oncologist, using the, 0-6 Skin Reaction Scale. Also weekly assessment of patient comfort, using Legacy's patient subjective pain rating, (0 no pain to 10 severe pain). Patients will keep track of their own pain and the time of application of the study gel. They will do this daily and write it on the calendar provided to them. A 5 question survey related to their comfort will be completed by the study nurse at the last visit. Outcomes would be measured by degree of skin reaction, discomfort, and cosmetic outcome. Breaks in treatment schedule, secondary to skin changes would be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Breast Cancer

* Radiation

Exclusion Criteria:

1. Post Mastectomy
2. Previous irradiation of the same breast
3. Pregnacy
4. Younger than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Reduction in skin damage | Start of radiation therapy until completion
  Skin reaction scale along with evaluation by radiation oncologist at weekly intervals from start of radiation therapy until completion of radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Johnson, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Health System, Portland, Oregon, United States

REFERENCES:
- [Result] Miko Enomoto T, Johnson T, Peterson N, Homer L, Walts D, Johnson N. Combination glutathione and anthocyanins as an alternative for skin care during external-beam radiation. Am J Surg. 2005 May;189(5):627-30; discussion 630-1. doi: 10.1016/j.amjsurg.2005.02.001. PMID 15862509
- See also: Related Info — http://www.legacyhealth.org